CLINICAL TRIAL: NCT06830564
Title: the Effect of the Low Dose Nalbuphine Versus Dexmedetomidine on the Prevention of Emergence Agitation After Sevoflurane Anaesthesia in Children Undergoing ENT Surgeries
Brief Title: Emergence Agitation of Sevoflurane in Pediatric
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FMASU MS127/2024
Record Dates: First submitted 2024-11-28; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Emergence Delirium
Keywords: Emergence delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Nalbuphine; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: paediatric patients undergoing ENT surgeries will be randomly assigned into one of the following groups using computer generated codes and opaque sealed envelopes:
  1. Group A will receive dexmedetomidine IV 0.5 μg/kg.
  2. Group B will receive nalbuphine IV 0 .1 mg /kg.
Who Masked: Participant, Care Provider, Investigator
Masking Description: prospective, randomized, double-blinded, comparative study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nalbuphine group (Active Comparator): We will give the patient before extubation by15 minute nalbuphine with dose 0.1 mg /kg and we will assess the emergence agitation by delirium score every 15 minutes for half an hour
  Interventions: Drug: we will give the patient 0.1 mg nalbuphine 15 min before the end of the procedure
- Dexmedetomidine group (Active Comparator): We will give the patient before extubation by 15 minute nalbuphine with dose 0.5 mic /kg and we will assess the emergence agitation by delirium score every 15 minutes for half an hour
  Interventions: Drug: we will give the patient 0.5 mg dexmedetomidine 15 min before the end of the procedure

INTERVENTIONS:
Drug: we will give the patient 0.1 mg nalbuphine 15 min before the end of the procedure — The study medications will be prepared by the local pharmacy as 10 ml syringes of nalbuphine IV that will be handled to the anesthesiologist in charge in OR room who will be blinded to the nature of the medications used, and study medications will be given 15 minutes before the end of surgical procedure and it will be given slowly for five minutes. . After extubation, patients will be taken to postanesthetic care unit . on arrival vital data will be measured. The anesthesiologist following up the patient will be blinded to the groups. The time of extubation will be defined as zero and after 15 minutes will be defined as one . Assessment of agitation will be done at time zero and time 1 and every fifteen minutes for 30 minutes using paediatric anaesthesia Emergence delirium scale (PAEDS)
  Arms: Nalbuphine group
Drug: we will give the patient 0.5 mg dexmedetomidine 15 min before the end of the procedure — The study medications will be prepared by the local pharmacy as 10 ml syringes of dexmedetomidine IV that will be handled to the anesthesiologist in charge in OR room who will be blinded to the nature of the medications used, and study medications will be given 15 minutes before the end of surgical procedure and it will be given slowly for five minutes. . After extubation, patients will be taken to postanesthetic care unit . on arrival vital data will be measured. The anesthesiologist following up the patient will be blinded to the groups. The time of extubation will be defined as zero and after 15 minutes will be defined as one . Assessment of agitation will be done at time zero and time 1 and every fifteen minutes for 30 minutes using pediatric anesthesia Emergence delirium scale (PAEDS) .
  Arms: Dexmedetomidine group

SUMMARY:
Low dose nalbuphine versus dexmedetomidine on prevention of emergence agitation in children

DETAILED DESCRIPTION:
The incidence of emergence agitation (EA) varies between 18% and 80.

EA occurs most frequently in preschool children during the early stage of emergence from anaesthesia .

It is considered a potentially serious postoperative complication that can result in physical harm and removal of intravenous catheters. As such, EA is a source of dissatisfaction for the parents of paediatric patients and their healthcare providers .

Sevoflurane is an inhalational anaesthetic used widely as a paediatric or outpatient anaesthesia due to its excellent hemodynamic stability and low blood solubility, which allows rapid induction and emergence from general anaesthesia, as well as control of the depth of anaesthesia. However, when sevoflurane is used alone it is associated with a higher incidence of emergence agitation in children. The rapid removal of residual anaesthetics due to low blood solubility of sevoflurane has been suggested to cause emergence agitation in some patients

Nalbuphine is a semi-synthetic, agonist antagonist opioid analgesic agent that acts as a partial agonist at kappa receptors and an antagonist at µ receptors, has minimal side effects, and exhibits a ceiling effect for respiratory depression .

Nalbuphine should effectively relieve postoperative pain and decrease the rate of EA in paediatric patients after sevoflurane anaesthesia.

Dexmedetomidine, a selective alpha 2 agonist, has been shown to reduce the incidence of postoperative agitation with sevoflurane anaesthesia .

Dexmedetomidine can affect the brain and spinal cord α 2-adrenergic receptor, inhibition of neural discharge to produce sedative, analgesic, and anxiolytic effects.

The Locus Coeruleus is a verified key part of the brain responsible for the regulation of arousal and sleep. Dexmedetomidine affects the brainstem locus coeruleus α 2-adrenergic receptors and produces sedative, hypnotic, and anxiolytic effects and it has also anesthetic-sparing effects without significant respiratory depression .

This study will be conducted to evaluate the effect of intravenous nalbuphine IV 0.1 mg/kg versus Dexmedetomidine IV 0.5 μg/kg on EA in paediatric patients undergoing ENT surgeries under sevoflurane anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age 4 - 10 years.
* Sex: male and female
* Patients with ASA classification I and II

Exclusion Criteria:

* Refusal of the caregiver to give written informed consent.
* History of allergy to the medications used in the study.
* psychiatric disorder.
* ASA classification III - IV.
* Fever, cough, asthma or upper respiratory tract infection.
* surgery more than 2 hours
* Hearing defect that limits communication.
* Neurological disorder .
* History of malignant hyperthermia.
* surgeries more than 2 hours.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
incidence of emergence agitation after sevoflurane anaesthesia | 6 months
  The aim of this study is to prevent 80% of emergence agitation of pediatric undergoing ENT surgeries using sevoflurane as inhalational anaesthesia . low dose nalbuphine versus dexmedetomidine

CONTACTS AND LOCATIONS:
Overall Officials: Madlin A selwanes, M.B.B.CH, Principal Investigator — anesthesia resident at Ain shames university
Locations (1):
- Ainshams University, Cairo, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all date should be shared once the study is published
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 6/2025
Access Criteria: Free